CLINICAL TRIAL: NCT05848115
Title: Understanding the Role of Bilevel Positive Airway Pressure (BiPAP) in Pediatric Acute Asthma Exacerbations: A Prospective, Randomized, Double Blind, Controlled Trial
Brief Title: BiPAP in Pediatric Moderate to Severe Asthma Randomized Control Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim Analysis showed futility for the primary outcome measure.
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-2338; 1R61HL158814-01A1 (NIH)
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Asthma in Children
Keywords: Pediatric Asthma; Asthma; Bi-level Positive Airway Pressure; BiPAP; Beta-Agonist
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BiPAP (Experimental): Patients randomized to the study group (BiPAP) will receive continuous nebulized albuterol through the FDA approved Respironics Trilogy BiPAP machine as per routine practice and institutional guidelines for albuterol dosing. Participants will receive BiPAP for four hours or until weaned off continuous beta-agonist therapy by the treating clinician.
  Interventions: Device: Bi-level Positive Airway Pressure
- Control (Sham Comparator): Patients randomized to the control group (sham BiPAP) will receive continuous nebulized albuterol through the same set-up as the study group and institutional guidelines for albuterol dosing. Participants will remain on sham BiPAP for four hours or until weaned off continuous beta-agonist therapy per the treating clinician.
  Interventions: Device: Sham Bi-level Positive Airway Pressure

INTERVENTIONS:
Device: Bi-level Positive Airway Pressure — An appropriately sized vented BiPAP face mask with a good seal will be applied and monitored by trained respiratory therapists. Patients will be started on an inspiratory peak airway pressure (IPAP) of 10 cm of water and expiratory positive airway pressure (EPAP) of 5 cm of water per Children's Hospital Colorado (CHCO) clinical pathway. BiPAP pressures will be titrated to effect per the treating physician, using assessment of physical examination, vitals, and asthma score per institutional clinical pathway. Study participants will remain on BiPAP for four hours or until weaned off continuous beta-agonist therapy by the treating clinician. After the four-hour intervention period, it is at the discretion of the treating clinician regarding the ongoing use of BiPAP or not.
  Other Names: BiPAP
  Arms: BiPAP
Device: Sham Bi-level Positive Airway Pressure — The sham BiPAP will have pressure attenuated using an orifice restrictor as described in previous double blinded studies using sham non-invasive ventilation. With this set-up pressures no greater than 2 cm of water have been documented at the location of the face mask. This will ensure that the patient is not receiving positive pressure with any effectiveness or deleterious effects. Study participants will remain on sham BiPAP for four hours or until weaned off continuous beta-agonist therapy by the treating clinician. After the four-hour intervention period, it is at the discretion of the treating clinician regarding the use of BiPAP or not.
  Other Names: Sham BiPAP
  Arms: Control

SUMMARY:
The goal of this clinical trial is to study if starting bi-level positive airway pressure (BiPAP), a mask that gives pressure to the lungs, works well for children in the emergency department with moderate to severe asthma attacks. The main questions it aims to answer are:

1. Whether initiation of BiPAP at the same time as continuous beta-agonist therapy (e.g., nebulized albuterol) will decrease how long children with moderate to severe asthma attacks need to receive continuous beta-agonist therapy.
2. Whether early BiPAP changes how the lungs function in children with asthma attacks.
3. Whether children receiving early BiPAP experience more issues or side effects than those children who do not.

All children will receive the usual treatment for asthma attacks; if they are still experiencing moderate to severe symptoms after the initial treatment, they will be asked to participate in the study. Participants will then wear a mask while they are receiving the continuous beta-agonist therapy. Some patients will receive BiPAP where pressure is given to the lungs and others will have a sham BiPAP mask where no pressure is given to the lungs. Study participants will wear the mask for 4 hours or until their treatment team feels they are ready to come off of the continuous beta-agonist therapy. Participants will receive more medications and decisions on going home or being admitted to the hospital will be decided as usual by their treatment team.

Researchers will compare BiPAP versus Control (Sham BiPAP) groups to see if there is a difference in how long continuous beta-agonist therapy is needed, how the lungs are functioning, and number or type of side effects.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 17 years of age (inclusive) presenting to the ED with an asthma exacerbation
* Prior diagnosis of asthma by a physician who prescribed asthma medications (beta-agonist and/or inhaled or oral steroids)
* PRAM score of 4 or greater after administration of first-line therapy (albuterol/ipratropium back to backs, corticosteroids, +/- oxygen) and need for continuous beta-agonist therapy after first-line therapy

Exclusion Criteria:

* Prior participation in the study
* Hypercapnic (PaCO2 > 60 mmHg) respiratory failure or need for invasive mechanical ventilation as determined by the treating physician
* Hypoxemic respiratory failure (SaO2 < 90% with fraction of inspired oxygen inspired oxygen fraction (FiO2) > 0.35)
* Presence of a tracheostomy or baseline noninvasive ventilation requirement
* Non-asthma causes of wheezing: foreign body, tracheomalacia, vocal cord dysfunction, pulmonary edema, uncorrected congenital heart disease, cystic fibrosis, anaphylaxis
* Absolute or relative contraindication to BiPAP: facial trauma, uncontrollable vomiting, hypotension for age, Glasgow Coma Score of 8 or less, drowsiness or confusion, known or clinical suspicion for pneumothorax, pneumomediastinum, or subcutaneous emphysema, pregnancy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Duration of Continuous Beta-Agonist Therapy | Through study completion, an average of 24 hours
  Number of hours until discontinuation of continuous beta-agonist therapy

SECONDARY OUTCOMES:
Change in Pediatric Respiratory Assessment Measure (PRAM) | At two and four hours after starting the intervention
  Change in Pediatric Respiratory Assessment Measure (PRAM) from baseline to two and four hours, minimum score of 0 and maximum score of 12, the higher the score the more severe the disease
Change in Respiratory Rate | At two and four hours after starting the intervention
  Change in respiratory rate in breaths per minute from baseline to two and four hours
Invasive Mechanical Ventilation | Four-hour study intervention
  Rate of participants requiring endotracheal intubation for invasive mechanical ventilation
Admission to Pediatric Intensive Care Unit (PICU) | Through entire hospitalization, an average of 72 hours
  Rate of admissions to the Pediatric Intensive Care Unit (PICU)
Total Length of Stay in Hospital | Through entire hospitalization, an average of 72 hours
  Total length of stay in hours in the Emergency Department (ED), Pediatric Intensive Care Unit (PICU), and hospital floor
Hospital Readmissions | 7 days from hospital discharge date
  Rate of hospital readmission within 7 days
Duration of Bilevel Positive Airway Pressure (BiPAP) | Through entire hospitalization, an average of 72 hours
  Duration in hours of BiPAP administration
Adverse Events | Four-hour study intervention
  Pneumothorax, pneumomediastinum, sub-cutaneous emphysema, hypotension, vomiting, aspiration, skin breakdown
Change in Pulse Oxygen Saturation | At 2 hour and 4 hours after starting the intervention
  Change in pulse oxygen saturation (range from 0 to 100%) from baseline to two and four hours
Change in Heart Rate | At 2 hour and 4 hours after starting the intervention
  Change in heart rate in beats per minute from baseline to two and four hours

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Wilson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.